CLINICAL TRIAL: NCT01026883
Title: Evaluation of a Novel Method for Hematocrit Level Determination
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. Priv. - Doz. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OPHT-290909
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Healthy
Keywords: hematocrit; layered resonant piezoelectric sensors
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy subjects (Other): Hematocrit level of each subject will be assessed by two different techniques
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — A venous blood sample will be taken (15 ml). Blood will be collected in 5 tubes. To avoid hematocrit variations due to the blood draw procedure, the first tube will be discarded. After that, the tourniquet which is used for venipuncture will be removed and 4 EDTA tubes (each 3 ml) will be filled with blood for hematocrit determination, one tube will be sent to the Department of Laboratory Medicine, and the other ones will be processed at the Department of Clinical Pharmacology.

SUMMARY:
The hematocrit level is defined as the ratio of plasma volume and red blood cell mass. Determination of this level is important for the diagnosis and follow-up of various hematological and renal disorders. In clinical practice, automated hematology analyzers are commonly used.

Recently, a new method for hematocrit level determination has been introduced which employs layered resonant piezoelectric sensors. In the present study this technique will be applied in blood samples of healthy subjects and compared to a standard laboratory method.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 18 and 80 years
* Men and women will be included in equal parts
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Symptoms of a clinically relevant illness in the 3 weeks before the study day
* Systemic treatment with anticoagulants
* Intake of any medication that could lead to spurious hematocrit values
* Presence of any medical condition that could lead to spurious hematocrit values
* Blood or plasma donation during the previous 3 weeks

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Correlation of hematocrit level determined by two different techniques | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhofer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Vienna, Austria